CLINICAL TRIAL: NCT05350085
Title: A Randomized Controlled Clinical Trial of Remimazolam Benzenesulfonate Usage in the Extraction of Impacted Wisdom Teeth
Brief Title: Remimazolam in the Extraction of Impacted Wisdom Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Anzhen Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RBEIWT2022
Record Dates: First submitted 2022-04-10; First posted 2022-04-27 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2022-04

CONDITIONS: Dental Anxiety; Sedation Complication; Anterograde Amnesia
MeSH Terms: conditions — Amnesia, Anterograde | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Group (Experimental): Use remimazolam as sedation.Sufficient sedation is defined as Ramsay Sedation score grade III.
  Interventions: Drug: Remimazolam besylate
- Midazolam Group (Active Comparator): Use midazolam as sedation.Sufficient sedation is defined as Ramsay Sedation score grade III.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remimazolam besylate — ① initial dose: use a micro injection pump to pump remimazolam at the rate of 50mg/h, and observe for 4 ~ 8 minutes until Ramsay Sedation grade III，then start dental operation ; ② Maintenance dose: maintain the pump speed at 5 ~ 10mg/h，adjust the pump dose to maintain the patient at Ramsay Sedation grade III. ③ Additional dose: During the operation, if the patient has body movement reaction or cannot cooperate with the dentist, local anesthetics shall be given as remedy. ④ After the operation, stop the microinjection pump.
  Arms: Remimazolam Group
Drug: Midazolam — ① initial dose: use a micro injection pump to pump remazolam at the rate of 30mg/h, and observe for 4 ~ 8 minutes until Ramsay Sedation grade III，then start dental operation; ② Maintenance dose: maintain the pump speed at 3 ~ 6mg/h，adjust the pump dose to maintain the patient at Ramsay Sedation grade III. ③ Additional dose: During the operation, if the patient has body movement reaction or cannot cooperate with the dentist, local anesthetics shall be given as remedy. ④ After the operation, stop the microinjection pump.
  Arms: Midazolam Group

SUMMARY:
Benzodiazepines, represented by midazolam, are often used for sedation in outpatient surgery in dentistry. However, midazolam has the problems of slow consciousness recovery and long recovery time, which brings trouble to the patients. Remimazolam is a new type of ultra short acting sedative anesthetic. Compared with other similar products, remimazolam has faster effect, rapid metabolism and has no accumulation, which may mean that compared with midazolam, remimazolam has a better clinical application prospect in dental outpatient surgery.

DETAILED DESCRIPTION:
The patients were randomly divided into midazolam group and remimazolam group. The onset time of drugs, postoperative recovery time, vital signs, anterograde amnesia and other complications were observed.

ELIGIBILITY:
Inclusion Criteria:

Consenting patients will be eligible if they:

1. Have mandibular impacted wisdom teeth that need to be extracted;
2. Have a body mass index (BMI) between 18.5 and 30 kg/m2;
3. Are aged between 18 and 60 years;
4. Have American Society of Anesthesiology (ASA) classification grade of I-II;
5. Have Modified Dental Anxiety Scale (MDAS) score > 15; and
6. Volunteered to accept intravenous sedation.

Exclusion Criteria:

Patients will be ineligible if they:

1. Are pregnant;
2. Experience respiratory infections, asthma attack or persistent state;
3. Have contraindications to anaesthesia or a previous abnormal surgical anaesthesia recovery history;
4. Have severe cardiopulmonary insufficiency;
5. Have preoperative blood pressure > 160/100 mmHg or diastolic blood pressure > 100 mmHg, or blood pressure < 90/60 mmHg;
6. Have a neuromuscular or mental disorder that renders them unable to communicate or cooperate effectively or sign informed consent;
7. Are suspected of abusing narcotic analgesics or sedatives;
8. Have a known allergy or contraindication to benzodiazepines; or
9. Have participated in other drug trials within 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Recovery time of complete alertness | During treatment in hospital, an expected average of 2 hours
  Calculated from the cessation of sedative injection with micro injection pump, the patients were scored with the modified observer's assessment of alertness/sedation scale (MOAA/S) every 1 minute, and the first minute with MOAA/S score = 5 for 3 consecutive times. MOAA/S score: Range from 5(Awake) to 1(Unresponsive).

SECONDARY OUTCOMES:
Anterograde amnesia duration | During treatment in hospital, an expected average of 2 hours
  Patients were given 3 different cards(including animals, fruits, vegetables, vehicles）at 0， 15，30，60 minutes after complete alertness（described at primary outcome). They were asked to recall them immediately and delayed(approximately 5 minutes after Immediate memory).
Interruption reasons during operation | During treatment in hospital, an expected average of 2 hours
  It includes chokes, hypoxia, continuous movement that makes treatment difficult, or other situations requiring suspension of operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant dat that underlie the results reported, after deidentification, including texts, tables, figures, and appendices, will be shared as supplementary material.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Jing Q, Wang W, Wu L, Wang L, Yuan B, Wang Y, Wang C, Liu L, Guan L, Yu R, Zhang Y, Sessler DI, Huang Y, Wan K, Pei L. A Comparison of the Effect of Remimazolam and Midazolam on Recovery and Preserved Memory Function for Patients with Dental Extraction Anxiety. Drug Des Devel Ther. 2025 Dec 30;19:11977-11987. doi: 10.2147/DDDT.S551322. eCollection 2025. PMID 41488759
- [Derived] Wang L, Jing Q, Pei L, Li M, Ruan X, Chen S, Zhang Y, Wan K, Huang Y. Efficacy of continuous intravenous remimazolam versus midazolam in the extraction of impacted wisdom teeth: protocol of a randomised controlled trial. BMJ Open. 2023 Apr 25;13(4):e067908. doi: 10.1136/bmjopen-2022-067908. PMID 37185197